CLINICAL TRIAL: NCT05580471
Title: A Randomized Control Study of 4DryField PH Anti-Adhesion Agent After Colorectal Surgery
Brief Title: A Randomized Control Study of Anti-Adhesion Agent After Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, Chief of colorectal surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202106033
Record Dates: First submitted 2022-10-09; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Adhesion
Keywords: Adhesion; post-operation; Colorectal surgery
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Use 4DryField
  One group use 4DryField before wound closure. One group do not use 4DryField before wound closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use 4DryField (Experimental): One group use 4DryField before wound closure.
  Interventions: Device: Use 4DryField
- Not Use 4DryField (No Intervention): One group do not use 4DryField before wound closure.

INTERVENTIONS:
Device: Use 4DryField — Patients randomly use 4DryField in Colorectal resection combined with temporary stomy before fascia closure. We observed the adhesion severity and adhesion extent when stomy closure.
  Arms: Use 4DryField

SUMMARY:
This project is to evaluate the difference of post-operation adhesion severity and adhesion area of patient received 4DryField after colorectal surgery.

DETAILED DESCRIPTION:
This proposal will investigate the effect of the newly anti-adhesive agent 4DryField. Stoma creation is common in complicated colorectal disease. Hartman procedure (End colostomy) is used in patients advanced rectal cancer or severe diverticulitis. Loop colostomy or ileostomy is used in patients need stool diversion for prevent leakage related infection.

4DryField is a powder consisting of sterile hydrophilic microparticles, which is anufactured from highly purified potato starch in a complex process. A unique starch-based medical device is 4DryField® PH (4DryField; PlantTec Medical GmbH, Germany) as it is the only product proven to provide hemostasis and prevent the formation of adhesions. In rat model, the 4DryField acheieve the significant adhesion prevention effectiveness. In gynecologic surgery, 4DryField showed effective adhesion prevention as confirmed at second look laparoscopy. The gel is easilier to applied in the uneven surface of pelvic cavity and peristomy area than other manufacture. The indication of adhesion prevention is approved by TFDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal resection and temporary stoma

Exclusion Criteria:

* - Pregnancy, child, psychiatric disorder, behavior disorder, and prisoner. And those patients can't follow the protocol

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-05 (Actual); Primary Completion 2024-09-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Adhesion severity | 0 days
  Adhesion severity was scored as grade 0 (no adhesion), grade I (filmy adhesion and blunt dissection), grade II (strong adhesion and sharp dissection), and grade III (very strong vascularized adhesion, sharp dissection, and damage barely preventable)
Adhesion extent | 0 days
  Adhesion area was scored as grade 0 (no adhesion), grade I (adhesion of less than one-third of the observational area), grade II (adhesion of one-third and two-thirds of the observational area), and grade III (adhesion of more than two-thirds of observational area ).

SECONDARY OUTCOMES:
Length of hospital stay | 7-14 days
  Number of days in hospital after surgery
Complication | 30 days
  Complications within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tungcheng Chang, PhD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan